CLINICAL TRIAL: NCT06647979
Title: An Adaptive Design Basket Trial of Hematopoietic Stem Cell BCL11A Enhancer Gene Editing for Severe β-Hemoglobinopathies
Brief Title: Hematopoietic Stem Cell BCL11A Enhancer Gene Editing for Severe β-Hemoglobinopathies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Bauer (Other)
Responsible Party: Sponsor-Investigator, Daniel Bauer, Associate Professor Pediatrics, Boston Children's Hospital, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCH-201
Record Dates: First submitted 2024-10-11; First posted 2024-10-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia (HbSS, or HbSβ-thalassemia0); Beta-Thalassemia; Transfusion Dependent Beta-Thalassaemia
Keywords: gene therapy; stem cell transplant; bone marrow transplant; autologous hematopoietic stem cell transplant; gene editing; hematopoietic stem cell transplant
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia | interventions — Sequence Analysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Sickle Cell Disease and Transfusion-Dependent Beta-Thalassemia (Experimental)
  Interventions: Biological: autologous bone marrow derived CD34+ HSPCs electroporated with BCL11A enhancer targeting Cas9 ribonucleoprotein; Device: Sequencing Assay for Variant rs114518452

INTERVENTIONS:
Biological: autologous bone marrow derived CD34+ HSPCs electroporated with BCL11A enhancer targeting Cas9 ribonucleoprotein — autologous bone marrow derived CD34+ HSPCs electroporated with BCL11A enhancer targeting Cas9 ribonucleoprotein
Device: Sequencing Assay for Variant rs114518452 — Device used to carry out the diagnostic testing for exclusion criteria number 12

SUMMARY:
A promising approach for the treatment of genetic diseases is called gene therapy. Gene therapy is a relatively new field of medicine that uses genetic material (mostly DNA) from the patient to treat his or her own disease. In gene therapy, the investigators introduce new genetic material in order to fix or replace a diseased gene, with the goal of curing the disease. The procedure is similar to a bone marrow transplant, in that the patient's malfunctioning blood stem cells are reduced or eliminated using chemotherapy, but it is different because instead of using a different person's (donor) blood stem cells for the transplant, the patient's own blood stem cells are given back after the new genetic material has been introduced into those cells. This approach has the advantage of eliminating any risk of Graft-Versus-Host Disease (GVHD), reducing the risk of graft rejection, and may also allow less chemotherapy to be utilized for the conditioning portion of the transplant procedure. The method used to fix or replace a diseased gene is called gene editing. A person's own cells are edited using a specialized biological medicine that has been formulated for use in human beings.

Fetal hemoglobin (HbF) is a healthy, non-sickling kind of hemoglobin. Investigators have recently discovered a gene called BCL11A that is very important in the control of fetal hemoglobin expression. Increasing the expression of this gene in sickle cell patients could increase the amount of fetal hemoglobin while simultaneously reducing the amount of sickle hemoglobin in their blood, and therefore potentially cure the condition.

DETAILED DESCRIPTION:
This is a non-randomized, single center, open-label, pilot safety and feasibility study involving a single infusion of autologous bone marrow derived CD34+ hematopoietic stem cells (HSPCs) electroporated with BCL11A enhancer targeting Cas9 ribonucleoprotein. Accrual will be a maximum of 14 evaluable subjects with sickle cell disease (SCD) or β-thalassemia. The study will enroll 7 evaluable subjects within each disease group: SCD and β-thalassemia. The study will have two strata within each diagnosis group.

SCD

Ages ≥18-40 years: Stratum 1a (n=3-7)

Ages ≥13-18 years: Stratum 2a (n=0-4)

β-thalassemia

Ages ≥18-40 years: Stratum 1b (n=3-7)

Ages ≥13-18 years: Stratum 2b (n=0-4)

After meeting eligibility criteria, patients will be enrolled. Patients with SCD will receive blood transfusions for a period of 3 months prior to hematopoietic stem cell collection, with a goal of achieving a Hemoglobin S (HbS) level of ≤ 30% by the time of mobilization. All patients will undergo peripheral stem cell mobilization and have their cells collected by apheresis. The collected cells of each subject will be split into 2 portions; one portion for gene editing, and one portion set aside as a back-up product in the event a rescue treatment is needed. Patients may undergo multiple rounds of collection if sufficient numbers of cells are not obtained with the first collection.

Patients will undergo a standard work-up for autologous bone marrow transplantation prior to proceeding with conditioning and infusion of their gene-edited cells. Patients will receive myeloablative conditioning with busulfan administered on days -5 to -2, prior to the infusion of edited cells. The edited cells will be infused intravenously.

Patients will be followed for 24 months after the infusion of their gene edited cells.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of either a) sickle cell disease with genotype HbSS, HbS/B0 thalassemia, HbSD, or HbSO, or b) transfusion-dependent β-thalassemia
2. Age 13-40 years.
3. Clinically severe disease, defined as: For sickle cell disease, the presence of one or more of the following clinical complications: i) Minimum of two episodes of acute chest syndrome (ACS) in the 2 years before study entry. ii) History of three or more episodes of severe pain events requiring a visit to a medical facility and treatment with parenteral opioids in the 2 years before study entry. For β-thalassemia patients: i) At least 100 mL/kg/year or 10 units/year of blood transfusions, on an annualized basis for the two years preceding enrollment.
4. Adequate hematologic parameters including:

   1. White blood cell (WBC) count within the range of 2.5 - 25.0 x 109 /L
   2. Platelet count within the range of 150 - 700 x 109 /L
5. Adequate organ function and performance status:

   1. Karnofsky performance status ≥70%
   2. Serum creatinine </=1.5 times the upper limit of normal for age, and calculated creatinine clearance or GFR </= 60 mL/min/1.73 m2.
   3. Direct bilirubin ≤ 2.0 mg/dL
   4. DLCO (corrected for hemoglobin), FEV1, FVC >50% of predicted
   5. Left ventricular ejection fraction >40% or shortening fraction >25%
6. For sickle cell patients: Failure of hydroxyurea therapy due to lack of clinical improvement, inability to tolerate due to side effects (e.g., myelosuppression, gastrointestinal symptoms, or hepatic enzyme elevations) or not clinically indicated (such as in a patient on a chronic transfusion regimen). Clinical criteria (per above) must be met despite taking hydroxyurea for greater than or equal to 6 months, unless not indicated or not tolerated. Patients taking hydroxyurea who still meet all inclusion criteria are eligible for the trial. Hydroxyurea should be discontinued when transfusions prior to gene therapy begin.
7. Confirmed sickle cell disease or β-thalassemia diagnosis by molecular genetic testing.
8. No HLA genotypically-identical related appropriate bone marrow donor available.
9. Parental/guardian/patient signed informed consent.
10. Willingness to return for follow-up for 15 years.

Exclusion Criteria:

1. Subjects who have concomitant condition or illness including, but not limited to:

   1. Uncontrolled infection, such as current febrile illness, infection requiring parenteral antibiotics, or systemic fungal infection.
   2. Active malignancy.
   3. Active complication of underlying hemoglobinopathy that would place the patient at unacceptable risk for participation, in the judgment of the Investigators.
   4. Major surgery in the past 30 days.
   5. Medical/psychiatric illness/social situations that would limit compliance with study requirements as determined by the treating physician.
2. Contraindication to administration of conditioning medication (busulfan).
3. Subjects who have undergone allogeneic or autologous hematopoietic stem cell transplant previously.
4. Either or both of the following findings on screening bone marrow aspirate/biopsy: a) diagnosis of myelodysplastic syndrome (MDS) based on morphology and/or cytogenetics (based on WHO definitions) or b) pathogenic mutation in any gene on the Rapid Heme Panel (RHP), a next-generation targeted sequencing clinical assay for hematologic malignancy associated mutations.
5. For SCD patients:

   1. Severe cerebral vasculopathy (defined by occlusion or stenosis in the circle of Willis; or presence of Moyamoya disease)
   2. Receiving a chronic transfusion regimen for primary or secondary stroke prophylaxis. (Note: patients with a history of abnormal transcranial Doppler (TCD) who have transitioned from transfusions to hydroxyurea for stroke prophylaxis are also not eligible for the study. Most recent TCD must be within one year of screening for patients up to 16 years old.)
   3. History of overt stroke or any neurologic event lasting > 24 hours. (Note: patients with imaging evidence of silent stroke but not on a chronic transfusion regimen are not excluded.)
6. Severe iron overload that is deemed to be grounds for exclusion based on the opinion of the Principal Investigator.
7. Known positive HIV serology or HIV nucleic acid testing, or positive serology for HCV, HBV, or HTLV.
8. Known acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on prior biopsy.
9. Receipt of an investigational study drug or procedure within 90 days of study enrollment.
10. Pregnancy, or breastfeeding in a postpartum female, or absence of adequate contraception for fertile subjects. Females of child-bearing potential must agree to use a medically acceptable method of birth control such as oral contraceptive, intrauterine device, barrier and spermicide, or contraceptive implant/injection from Screening through at least 6 months after drug product infusion. Male subjects must agree to use effective contraception (including condoms) from Screening through at least 6 months after drug product infusion.
11. An assessment by the Investigators that the subject will not comply with the study procedures outlined in the study protocol, or that, as determined by the investigators and/or transplant physician, the subject has any other condition rendering the subject ineligible for HSCT or other study procedures.
12. Patients carrying at least one cytosine (C) alternate allele at the SNP site rs114518452, chr2:210530659-210530659 (GRCh38/hg38), where guanine (G) is the reference allele.

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Primary engraftment | 42 days
  Successful hematopoietic reconstitution after conditioning (defined by absolute neutrophil count (ANC) greater than or equal to 0.5 x 10^9 /L for three consecutive days without growth factor support), achieved by day 42 after day 0 of stem cell infusion (i.e., "primary engraftment").

SECONDARY OUTCOMES:
Hemoglobin | 24 months
  Total hemoglobin (in g/dL), hemoglobin fractions (A, F, and S in g/dL), percent HbF, and percent F cells
Platelet Engraftment | 42 days
  Platelet engraftment (defined as platelet count ≥20,000/L without transfusion for 7 days by day +42 after stem cell infusion)
Severe vaso-occlusive crises (for sickle cell disease (SCD) patients) | 24 months
  Change from baseline in incidence of severe vaso-occlusive crises (requiring emergency department visit or hospital admission)
Acute chest syndrome (for sickle cell disease (SCD) patients) | 24 months
  Change from baseline in incidence of acute chest syndrome
Stroke (for sickle cell disease (SCD) patients) | 24 months
  Change from baseline in incidence of stroke
Splenic sequestration (for sickle cell disease (SCD) patients) | 24 months
  Change from baseline in incidence of splenic sequestration
Transfusion requirement (for sickle cell disease (SCD) patients) | 24 months
  Change from baseline in transfusion requirement (in mL/kg) after day +100 post infusion
Reticulocyte count (for sickle cell disease (SCD) patients) | 24 months
  Change from baseline reticulocyte count
Bilirubin (for sickle cell disease (SCD) patients) | 24 months
  Change from baseline bilirubin
Lactate dehydrogenase (LDH) (for sickle cell disease (SCD) patients) | 24 months
  Change from baseline lactate dehydrogenase (LDH)
Quality of Life | 24 months
  Quality of life, assessed by administration of the PedsQL survey tool to the patient (or parents of young children) for subjects under 18 years old, and by administration of the SF-36 survey tool for adult subjects
Safety Outcome: Death | 24 months
  Occurrence of death
Safety Outcome: Malignancy, abnormal bone marrow cytogenetics, or myelodysplasia | 24 months
  Occurrence of malignancy, abnormal bone marrow cytogenetics, or myelodysplasia
Safety Outcome: Serious adverse events | 24 months
  Number of serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No